CLINICAL TRIAL: NCT07338058
Title: Effect of Fragmented Exercise Snacks on Mobile Phone Addiction and Psychophysical Health in Adolescents: A Randomized Controlled Trial
Brief Title: High-Intensity Exercise Snacks for Reducing Mobile Phone Addiction in Adolescents
Acronym: ES-MPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Responsible Party: Principal Investigator, Ma Ruisi, Lecturer, School of Physical Education, Jinan University, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBRE-25-0472; SBRE-25-0472 (Other: Survey and Behavioural Research Ethics Committee of The Chinese University of Hong Kong)
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Smartphone Addiction; Sedentary Behaviors; Adolescent Behavior
Keywords: Exercise Snacks; High-Intensity Interval Training; Fragmented Exercise; Self-Control; Digital Health
MeSH Terms: conditions — Internet Addiction Disorder; Sedentary Behavior; Adolescent Behavior; Self-Control

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with a parallel group design. Eligible participants are randomly assigned to either the Exercise Snacks intervention group or the control group in a 1:1 allocation ratio. Randomization is performed using computer-generated random number sequences to ensure equal probability of assignment.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the behavioral intervention (exercise training), it is not possible to blind the participants or the instructors to the group allocation. However, outcome assessors and data analysts are blinded to the group assignment to minimize detection and reporting bias. All data will be coded, and the statistical analysis will be conducted without knowledge of group identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Snacks Group (Experimental): Participants in this group follow a 5-month structured "Exercise Snacks" protocol. The intervention consists of daily short bursts of high-intensity exercise (e.g., 1-minute sprints, squats) performed during school breaks, supplemented by weekly collective HIIT sessions. The program progresses through adaptation, enhancement, and consolidation phases.
  Interventions: Behavioral: Exercise Snacks Protocol
- Control Group (No Intervention): Participants in this group are instructed to maintain their usual daily campus life and academic routines without altering their existing physical activity habits. They do not participate in the structured exercise snacks program during the study period.

INTERVENTIONS:
Behavioral: Exercise Snacks Protocol — The intervention consists of a structured 5-month "Exercise Snacks" program. Participants perform "snacks"-defined as isolated bouts of vigorous-intensity physical activity (<2 min)-distributed 3-4 times throughout the school day during breaks.
  Content: The regimen includes "Sprint Snacks" (e.g., stair climbing, high knees) and "Strength Snacks" (e.g., squats, push-ups). Intensity: Participants are instructed to reach a subjective effort level of Borg RPE > 14 (Somewhat Hard to Hard). Progression: The program follows a phased approach:
  Adaptation (Month 1): Focus on habit formation and movement quality.
  Enhancement (Months 2-3): Increased frequency and inclusion of weekly collective HIIT sessions.
  Consolidation (Months 4-5): Integration of cognitive-behavioral guidance to replace mobile phone usage habits.
  Other Names: Fragmented High-Intensity Exercise
  Arms: Exercise Snacks Group

SUMMARY:
This study is a randomized controlled trial (RCT) designed to evaluate the long-term effectiveness of "Exercise Snacks" (fragmented, high-intensity bouts of exercise) in reducing mobile phone addiction among adolescents.

Participants will be randomly assigned to either an intervention group or a control group. The intervention spans 5 months and is followed by a 1-month follow-up period (Month 6). The intervention group will perform short bursts of exercise (e.g., 1-minute sprints, squats) multiple times daily during school breaks. The program is divided into three progressive phases: adaptation, enhancement, and consolidation. The study aims to determine whether this sustained "snack-style" exercise regimen can significantly lower mobile phone addiction scores, improve physical fitness, and enhance psychological traits such as self-control and resilience over a semester-long period.

DETAILED DESCRIPTION:
Background and Rationale: Adolescents face increasing risks of mobile phone addiction, which is associated with sedentary behavior. "Exercise Snacks"-isolated bouts of vigorous exercise performed periodically throughout the day-offer a time-efficient solution. This study applies the COMB model and Self-Determination Theory to a long-term, semester-based intervention.

Study Design: This is a single-blind, randomized controlled trial conducted over a 6-month period (5 months of intervention + 1 month of follow-up).

Intervention Protocol: The intervention group follows a progressive "Exercise Snacks" program:

Adaptation Phase (Month 1 / Weeks 1-4): Focus on habit formation. Participants perform "Sprint Snacks" (e.g., stair climbing) 3 times daily and "Strength Snacks" (e.g., squats) 2 times weekly. Intensity is monitored to ensure safety and correct posture.

Enhancement Phase (Months 2-3 / Weeks 5-12): Focus on physiological adaptation. Frequency increases to 4 daily Sprint Snacks and 3 weekly Strength Snacks. A weekly collective High-Intensity Interval Training (HIIT) session is introduced to maximize cardiorespiratory benefits.

Consolidation Phase (Months 4-5 / Weeks 13-20): Focus on psychological integration. Daily snacks continue. Collective HIIT sessions increase to twice weekly. A cognitive-behavioral guidance component is added (bi-weekly) to help students identify phone use triggers and internalize healthy behaviors.

Follow-up Phase (Month 6 / Weeks 21-24): The structured intervention ceases. Participants are encouraged to maintain self-guided exercise. Final assessments are conducted at the end of Month 6 to evaluate the retention of intervention effects and any "rebound" in mobile phone addiction.

Outcome Measures: The primary outcome is Mobile Phone Addiction (SAS-SV), assessed at baseline, Month 3, Month 5 (post-intervention), and Month 6 (follow-up). Secondary outcomes include physical activity levels (PARS-3 and wearables), self-control (BSCS), resilience (RSCA), and mental health status.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 12-18 years enrolled in the participating middle/high school.
2. Owner of a smartphone with daily usage time > 2 hours.
3. Score on the Smartphone Addiction Scale-Short Version (SAS-SV) indicating a risk of addiction (e.g., score > 31 for males, > 33 for females).
4. Physically capable of participating in high-intensity exercise (PAR-Q screening negative).
5. Provided written informed consent (from both student and guardian).

Exclusion Criteria:

1. Diagnosed with severe physical disabilities or cardiovascular diseases that contraindicate high-intensity exercise (e.g., congenital heart disease).
2. Currently participating in other professional sports training or weight loss programs.
3. Diagnosed with severe psychiatric disorders (e.g., severe depression, schizophrenia) requiring medication.
4. Taking medications that affect heart rate or cognitive function.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mobile Phone Addiction Severity (assessed by SAS-SV) | Baseline, Month 3, Month 5, and Month 6
  The severity of mobile phone addiction is measured using the Smartphone Addiction Scale-Short Version (SAS-SV). This self-report scale consists of 10 items. Each item is rated on a 6-point Likert scale ranging from 1 ("Strongly Disagree") to 6 ("Strongly Agree"). The total score is calculated by summing the scores of all 10 items, resulting in a range from 10 to 60. Higher scores indicate a higher level of mobile phone addiction risk.

SECONDARY OUTCOMES:
Psychological Resilience(CD-RISC-10 Score) | Baseline, Month 3,Month 5, and Month 6
  10 items, 0-4 scale. Range 0-40. Higher scores indicate greater resilience.
Self-Control Capacity (BSCS Score) | Baseline, Month 3, Month 5, and Month 6.
  13 items, 1-5 scale. Range 13-65. Higher scores indicate better self-control.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Si Ma, Principal Investigator — Jinan University
Locations (1):
- School of Physical Education, Jinan University, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the article will be shared. This includes the text, tables, figures, and appendices. Data will be anonymized to protect participant privacy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months following article publication and ending 5 years following article publication.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal for meta-analysis or verification purposes. Proposals should be directed to the Principal Investigator at penny@link.cuhk.edu.hk. To gain access, data requestors will need to sign a data access agreement.